CLINICAL TRIAL: NCT02881580
Title: Risk Factors for Proximal Junctional Kyphosis Assessment After Spinal Instrumentation
Acronym: CYPHORACHI
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CYPHORACHI
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2016-08

CONDITIONS: Spinal Deformity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention : descriptive study

SUMMARY:
The surgical management of spinal deformities especially in adults is complex. The conventional surgical treatment of these deformations is a scope arthrodesis of the spine. The quality of the result depends on many variables such as the choice of the vertebrae to fuse, location and the number of implants, the type of material used or the type of correction maneuver used.

All these variables affect the surgical outcome and may be involved as a modifiable risk factor for possible postoperative complications. The study proposes to focus on the junctional kyphosis postoperative proximal (CJP or Proximal Junctional Kyphosis: PJK). Their prevalence in adults ranges from 20% to 43% depending on the series.

The radiographic definition of CJP's kyphosis with an angle> 10 ° measured from the lower plate of the proximal instrumented vertebra to the upper plate of the adjacent vertebra proximal not instrumented; this measure is being compared to the pre operative data.

Either the CJP are asymptomatic and do not require revision surgery either they are and thereby generate a revision surgery.

Several factors may potentially influence the development of the CJP. Among them, age, preoperative comorbidities, obesity, osteoporosis, lesions of the posterior elements, hybrid instrumentation, correction forces applied during surgery, sagittal balance pre and post operative degeneration joint capsules, etc. There are few studies on the identification and analysis of these risk factors; literature gives only single-center studies on small samples with a single surgical procedure. Review articles describe the incidence and risk factors of the CJP. However, the pathophysiological mechanisms of the CJP are still controversial to this day.

The aim of this study is to determine the incidence of occurrence of postoperative kyphosis proximal junctional and identify risk factors for developing this major complication of a multicenter population of scoliosis operated an extensive fusion.

DETAILED DESCRIPTION:
objectives:

Determine on a homogenous population of scoliosis operated for an extended fusion of 4 or more vertebrae:

* the incidence of proximal junctional kyphosis
* Modifiable risk factors and non modifiable of occurrence of CJP.
* the rate of CJP leading to revision surgery and the surgical recovery factors.

Methodology :

This is a multicenter retrospective cohort enrolling in Chapter X of the Data Protection Act and provides, as part of this research, the collection of individual data for evaluation of care and prevention practices with authorization request to the CNIL; the opinion of CCTIRS is not required in this case.

This study concerns the data of patients operated with the techniques mentioned in addition with more than 6 months back.

Patients are aware of the potential use of their data in their files for medical research through oral information provided by the doctor at the signing by the patient's consent related to the surgery and most recently contained in the Home booklet setting for patients.

Time study: 8 months Acquisition of data: KEOPS Database (declared to CNIL)

List of data to collect:

* Epidemiological data and conventional clinics.
* Background
* Questionnaires and functional scores when available. (Some patients filled out questionnaires in the prospective follow-up of results and signed an agreement on their inclusion in the Keops database.)
* Operating data
* X-rays of the entire spine from the front and side: pre-operative, post-operative and at last follow.

ELIGIBILITY:
Inclusion Criteria:

* age over 40 years
* Decline minimum 6 months
* Scoliosis degenerative etiology, neurological and idiopathic.
* segmental instrumentation over 3 levels (4 vertebrae) in the lumbar area.
* Patients operated on for the 1st time.

Exclusion Criteria:

* Lumbar spinal surgery or history of chest instrumented
* Etiology post traumatic tumor
* non-segmental instrumentation (Harrington type)
* segmental instrumentation on less than 3 levels.
* Pre and unreadable or missing postoperative radiograph
* Decline <6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Saint Joseph Hospital
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of proximal junctional kyphosis | Day 1

SECONDARY OUTCOMES:
Number of proximal junctional kyphosis leading to revision surgery and the surgical recovery factors. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume P RIOUALLON, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided